CLINICAL TRIAL: NCT00256425
Title: Cognitive Rehabilitation of Glioma Patients: a Prospective, Randomized Study
Brief Title: Cognitive Rehabilitation of Glioma Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: Dutch Cancer Society (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UU 2003-2783
Record Dates: First submitted 2005-11-18; First posted 2005-11-21 (Estimated); Last update posted 2008-03-21 (Estimated); Status verified 2007-07

CONDITIONS: Glioma; Cognition Disorders
Keywords: glioma; brain tumor; cognit; neuropsycholog; attention; memory; executive function; rehabilitation; remediation; training
MeSH Terms: conditions — Glioma; Cognition Disorders; Brain Neoplasms | interventions — Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Cognitive rehabilitation

SUMMARY:
The purpose of this study is to determine whether cognitive rehabilitation is effective in patients with gliomas (brain tumour), by comparing direct and follow-up neuropsychological functioning and quality of life of the experimental group to the control group.

DETAILED DESCRIPTION:
The majority of patients with (low-grade) glioma exhibit cognitive symptoms and objective deficits, which have a sustained, negative impact on daily functioning and quality of life.

Adult patients with a low-grade glioma, either histologically proven, or suspected (1), as well as adult anaplastic glioma patients with favorable prognostic factors (2), who are clinically stable for at least 6 months, will be recruited from 9 hospitals in the Netherlands. Consenting patients with both subjective cognitive symptoms and objective deficits will be randomized to either the cognitive rehabilitation program (N = 75) or a "waiting-list" control group (N = 75). Upon completion of the study, those patients assigned to the control group will be given the opportunity to undergo the cognitive rehabilitation program.

The cognitive rehabilitation program incorporates both retraining of impaired cognitive functions, and teaching of compensatory strategies. Rehabilitation will be directed towards attention, memory and executive functioning. The intervention will consist of 6 weekly, individual, 2-hour sessions plus two hours of homework.

To evaluate the efficacy of the rehabilitation program, objective neuropsychological functioning, self-reported cognitive symptoms and health-related quality of life will be assessed before rehabilitation, directly following rehabilitation, and at 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with a histologically proven low-grade glioma or presumed (i.e., suspected) low-grade glioma based on both clinical and MR imaging feature, and
* adult patients with an anaplastic glioma (anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic oligo-astrocytoma) under age 50 and with good performance status (KPS > 70);
* who are clinically stable for a minimum of 6 months prior to study entry (as determined by recent CT or MRI imaging) and no anti-tumor treatment during that period of time (i.e., surgery, radiotherapy, chemotherapy, corticosteroids);
* who report at least one symptom of impaired cognitive functioning based on a standardized self-report questionnaire, administered by researcher;
* and who meet criteria for neuropsychological impairment based on objective test results (assessed by researcher).

Exclusion Criteria:

* lack of basic proficiency in Dutch;
* IQ below 85;
* severe reading problems;
* an additional (history of) neurological or psychiatric disorder;
* participating in a concurrent study in which neuropsychological testing and/or health-related quality of life assessments are involved

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2003-10; Study Completion 2007-09 (Estimated)

PRIMARY OUTCOMES:
neuropsychological measures of attention (test scores) | baseline, immediately after 6 weeks and at 6-month follow-up

SECONDARY OUTCOMES:
neuropsychological measures of memory and executive functioning (test scores) | baseline, immediately after 6 weeks and at 6-month follow-up
subjective neuropsychological functioning (questionnaires) | baseline, immediately after 6 weeks and at 6-month follow-up
quality of life (questionnaires) | baseline, immediately after 6 weeks and at 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Martin JB Taphoorn, MD, PhD, Principal Investigator — Medical Center Haaglanden; Neil K Aaronson, PhD, Principal Investigator — The Netherlands Cancer Institute; Margriet M Sitskoorn, PhD, Principal Investigator — UMC Utrecht
Locations (9):
- Netherlands (9):
  - VU Medical Center, Amsterdam
  - Netherlands Cancer Institute, Amsterdam
  - UMC Groningen, Groningen
  - AZ Maastricht, Maastricht
  - UMC St Radboud, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - Medical Center Haaglanden, The Hague
  - Sint Elisabeth Hospital, Tilburg
  - University Medical Center Utrecht, Utrecht

REFERENCES:
- [Background] Klein M, Heimans JJ, Aaronson NK, van der Ploeg HM, Grit J, Muller M, Postma TJ, Mooij JJ, Boerman RH, Beute GN, Ossenkoppele GJ, van Imhoff GW, Dekker AW, Jolles J, Slotman BJ, Struikmans H, Taphoorn MJ. Effect of radiotherapy and other treatment-related factors on mid-term to long-term cognitive sequelae in low-grade gliomas: a comparative study. Lancet. 2002 Nov 2;360(9343):1361-8. doi: 10.1016/s0140-6736(02)11398-5. PMID 12423981
- [Background] Taphoorn MJ, Klein M. Cognitive deficits in adult patients with brain tumours. Lancet Neurol. 2004 Mar;3(3):159-68. doi: 10.1016/S1474-4422(04)00680-5. PMID 14980531